CLINICAL TRIAL: NCT01562834
Title: Randomized Cross Over Double Blind Versus Placebo Trial Followed by an Open Phase Studying Effect of Norditropin® on Left Ventricular Mass of Growth Hormone Deficient Adult Patients
Brief Title: Effect of Somatropin on Left Ventricular Mass in Growth Hormone Deficient Adult Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GHDADULT/F/1/F
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Somatropin (Experimental)
  Interventions: Drug: somatropin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: somatropin — Initial dosage 0.5 IU/day, injected subcutaneously (s.c., under the skin) once daily. Dosage will be adjusted monthly depending on clinical safety up to a maximum dose of 3 IU/day. Subjects are treated for six months (randomised trial period) followed by an 12-month open-label trial period with somatropin.
  Arms: Somatropin
Drug: placebo — Initial dosage 0.5 IU/day, injected subcutaneously (s.c., under the skin) once daily. Dosage will be adjusted monthly depending on clinical safety up to a maximum dose of 3 IU/day. Subjects are treated for six months. After treatment in the randomised trial period, placebo will be discontinued.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess the effect of somatropin (Norditropin®) replacement therapy on the left ventricular mass of adult patients with a growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Childhood or adult onset growth hormone deficiency (GHD)
* GHD evidenced by two stimulation tests
* Duration of GHD at least 5 years
* Other hormone deficiencies associated with growth hormone deficiency

Exclusion Criteria:

* Pregnancy or pregnancy desired during the suggested duration of the study
* Personal history of colonic polyp or family history of colonic polyposis
* Known insulin-dependent or non-insulin-dependent diabetes
* Cardiovascular disease, left ventricular hypertrophy from other aetiology, recent auricular or ventricular arrhythmia, history of vascularisation by aortocoronary bypass significative mitral or aortic valvular disease, preexcitation syndrome, auriculoventricular conduction delay, bradycardia-tachycardia syndrome, left ventricular mass interfering treatment
* BMI (Body Mass Index) at least 30
* Growth hormone treatment during the 24 months prior to inclusion, history of treatment with extractive pituitary growth hormone, allergy or suspected allergy to somatropin therapy
* Patient who has participated in a different clinical study within the past two months
* Any condition which, in the opinion of the Investigator or the Scientific Committee, may interfere with successful implementation of the study
* Notion of breast cancer for the mother or the sister

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 1998-10-21 (Actual); Primary Completion 2002-12-01 (Actual); Study Completion 2002-12-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass measured with ultrasonography

SECONDARY OUTCOMES:
Ventricular function indices assessed by cardiac ultrasonography
Bone mineral density and body composition assessed by DEXA (Dual Energy X-Ray Absorptiometry)
Quality of life using EQ5D (European Quality of Life 5 Dimensions) scales
IGF-I (Insulin-Like Growth Factor I) concentration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (20):
- France (20):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Boisguillaume
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Lorient
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Marseille Cédex 05
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Reims
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Tours
  - Novo Nordisk Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com